CLINICAL TRIAL: NCT04151563
Title: A Phase 1/2, Randomized Study Evaluating Multiple Nivolumab Combination Therapies in Patients With Stage IV or Recurrent Non-Small Cell Lung Cancer (NSCLC) After Failure of Platinum-Based Chemotherapy and Anti-PD-1 (L)1 Immunotherapy
Brief Title: A Clinical Study Evaluating Nivolumab-containing Treatments in Patients With Advanced Non-small Cell Lung Cancer After Failing Previous PD-1/(L)1 Therapy and Chemotherapy
Acronym: CheckMate 79X
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Clovis Oncology, Inc. (Industry); Exelixis (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-79X; 2018-004283-65 (EudraCT Number)
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Ipilimumab; cabozantinib; Docetaxel; Ramucirumab; E-3810

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A: cabozantinib + nivolumab + ipilimumab (Experimental)
  Interventions: Biological: nivolumab; Biological: ipilimumab; Drug: cabozantinib
- Arm B: cabozantinib + nivolumab (Experimental)
  Interventions: Biological: nivolumab; Drug: cabozantinib
- Arm C: nivolumab + ramucirumab + docetaxel (Experimental)
  Interventions: Biological: nivolumab; Biological: docetaxel; Biological: ramucirumab
- Arm D: lucitanib + nivolumab (Experimental)
  Interventions: Biological: nivolumab; Drug: lucitanib
- Arm E: nivolumab + docetaxel (Experimental)
  Interventions: Biological: nivolumab; Biological: docetaxel
- Arm F: docetaxel (Active Comparator)
  Interventions: Biological: docetaxel

INTERVENTIONS:
Biological: nivolumab — Specified dose on Specified days
  Other Names: OPDIVO; BMS-936558
  Arms: Arm A: cabozantinib + nivolumab + ipilimumab; Arm B: cabozantinib + nivolumab; Arm C: nivolumab + ramucirumab + docetaxel; Arm D: lucitanib + nivolumab; Arm E: nivolumab + docetaxel
Biological: ipilimumab — Specified dose on Specified days
  Other Names: YERVOY
  Arms: Arm A: cabozantinib + nivolumab + ipilimumab
Drug: cabozantinib — Specified dose on Specified days
  Other Names: CABOMETYX
  Arms: Arm A: cabozantinib + nivolumab + ipilimumab; Arm B: cabozantinib + nivolumab
Biological: docetaxel — Specified dose on Specified days
  Arms: Arm C: nivolumab + ramucirumab + docetaxel; Arm E: nivolumab + docetaxel; Arm F: docetaxel
Biological: ramucirumab — Specified dose on Specified days
  Other Names: CYRAMZA
  Arms: Arm C: nivolumab + ramucirumab + docetaxel
Drug: lucitanib — Specified dose on Specified days
  Other Names: CO-3810
  Arms: Arm D: lucitanib + nivolumab

SUMMARY:
This study is for participants with Non-small Cell Lung Cancer that has spread or has reoccurred after failure of Chemotherapy and Immunotherapy

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria

* Histologically or cytologically-documented Stage IV A/B non-small cell lung Cancer, stage IIIB/C disease failed concurrent chemoRT.
* ECOG Performance Status of ≤ 1.
* Radiologically-documented disease progression on one anti-PD-1/anti-PD-L1 therapy and one platinum-based doublet regimen given either concurrently or sequentially within 90 days after the last dose of anti-PD-(L)1.
* All participants must have tumor tissue submitted prior to randomization, either a recent archival sample obtained on/after the date of disease progression of the last prior anticancer therapy and within 3 months prior to enrollment, or a fresh biopsy obtained during the screening period.
* Prior toxicities must have resolved to grade ≤1.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test and must not be breastfeeding.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception. In addition, male participants must be willing to refrain from sperm donation during this time and must agree to follow instructions for method(s) of contraception. Azoospermic males are exempt from contraceptive requirements as well as WOCBP who are continuously not heterosexually active, however, a pregnancy test will still be required.

Exclusion Criteria

* Prior treatment with Docetaxel.
* Untreated CNS metastases, carcinomatous meningitis or leptomeningeal metastases.
* Any tumor invading the Superior Vena Cava other blood vessel, GI Tract or Trachea.
* EGFR mutations, ALK translocations, ROS1 translocations which are sensitive to inhibitor therapy.
* History of cerebrovascular accident and coagulation disorders.
* Participants with interstitial lung disease, history of cerebrovascular accident or history of abdominal fistula, gastrointestinal perforation, bowel obstruction, intra-abdominal abscess or grade 3-4 bleeding event within 6 months prior to randomization.
* Known toxicity on prior checkpoint inhibitor treatment.
* Participants who received more than one line of anti- PD-1/PD-L1 treatment.
* Participants who received previous CTLA-4 inhibitor treatment.
* Participants with known BRAF V600E mutation which are sensitive to available targeted inhibitor therapy are excluded.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2023-12-17 (Estimated); Study Completion 2026-05-13 (Estimated)

PRIMARY OUTCOMES:
Overall Reponse Rate (ORR) using RECIST 1.1 per Blinded Independent Central Review (BICR) assessment | approximately 33 months

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 Years
Duration of Response (DOR) by BICR using RECIST 1.1 | approximately 33 months
Progression-Free Survival (PFS) by BICR using RECIST 1.1 | Up to 5 Years
Incidence of Adverse Events (AEs) | Up to 5 Years
Incidence of Serious Adverse Events (SAEs) | Up to 5 Years
Incidence of Select AEs | Up to 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (22):
- Local Institution, Detroit, Michigan, United States
- Argentina (4):
  - Local Institution, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution, Buenos Aires, Distrito Federal
  - Local Institution, Caba, Distrito Federal
  - Local Institution, Capital, Distrito Federal
- Belgium (3):
  - Local Institution, Charleroi
  - Local Institution, Gilly
  - Local Institution, Leuven
- Local Institution, Copenhagen Ø, Denmark
- Greece (2):
  - Local Institution, Athens
  - Local Institution, Neo Faliro
- Mexico (4):
  - Local Institution, Torreón, Coahuila
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Puebla City, Puebla
- Netherlands (2):
  - Local Institution, Amsterdam
  - Local Institution, Rotterdam
- Local Institution, Oslo, Norway
- Poland (2):
  - Local Institution, Warsaw, Masovian Voivodeship
  - Local Institution, Krakow
- Romania (2):
  - Local Institution, Craiova
  - Local Institution, Timișoara

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm